CLINICAL TRIAL: NCT07339475
Title: Evaluation of Femoral Vein Diameter to Predict Intraoperative Hypotension in Geriatric Patients Undergoing Orthopedic Surgery Under Spinal Anesthesia: A Prospective Observational Study
Brief Title: Femoral Vein Diameter to Predict Intraoperative Hypotension in Geriatric Patients Undergoing Orthopedic Surgery Under Spinal Anesthesia
Status: Recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hebatallah Salah Abdelhamid, Lecturer of Anesthesia, Surgical Critical Care and Pain Management Department, Faculty of Medicine, Cairo University, Cairo, Egypt., Cairo University
Other Study IDs: MS-640-2025
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Femoral Vein Diameter; Intraoperative Hypotension; Orthopedic Surgery; Spinal Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Patients undergoing elective lower-limb orthopedic surgery under spinal anesthesia
  Interventions: Other: Measurement of Femoral Vein Diameter

INTERVENTIONS:
Other: Measurement of Femoral Vein Diameter — The transverse diameter of the right common femoral vein (RCFV) will be recorded 1 cm proximal to the junction with the great saphenous vein, at end-expiration.

SUMMARY:
The study aims to assess whether the transverse diameter of the right common femoral vein (RCFV) in the inguinal region could reflect the degree of post-spinal hypotension during elective orthopedic surgery.

DETAILED DESCRIPTION:
Spinal anesthesia is commonly used in orthopedic procedures but often results in hypotension, particularly in elderly patients due to reduced cardiovascular reserve and impaired autonomic function.

Ultrasound measurement of the right common femoral vein (RCFV) diameter has recently been proposed as a simple, non-invasive marker of intravascular volume status and a potential predictor of spinal anesthesia induced hypotension. To date, most evidence comes from obstetric populations undergoing cesarean delivery, limiting its applicability in other high-risk groups.

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years.
* American Society of Anesthesiologists (ASA) physical state I-II.
* Body mass index (BMI) ≤35 kg/m². Patients above this value will be excluded because obesity may cause technical difficulty and poor image quality in femoral vein ultrasound assessment.
* Elective lower-limb orthopedic surgery under spinal anesthesia.

Exclusion Criteria:

* Patients refusing to participate.
* History of psychiatric illness or seizures.
* Absolute contraindications to spinal anesthesia: infection at the puncture site, severe coagulopathy/anticoagulation [defined as platelet count <75,000/µL, International Normalized Ratio (INR) >1.5, Activated Partial Thromboplastin Time (aPTT) >1.5 times control, or the use of anticoagulants such as warfarin, heparin, low molecular weight heparin, or direct oral anticoagulants within the recommended safety interval for neuraxial anesthesia], severe hypovolemia, increased intracranial pressure, or known allergy to local anesthetics.
* Severe cardiac disease, including left ventricular ejection fraction <30%, Severe valvular heart disease (e.g., critical aortic stenosis), clinically significant arrhythmias (atrial fibrillation with uncontrolled ventricular rate >120 bpm, frequent ventricular ectopy or sustained ventricular tachyarrhythmia) and congestive heart failure such as New York Heart Association (NYHA) class III-IV.
* Severe uncontrolled hypertension, defined as persistent mean arterial pressure (MAP) ≥120 mmHg or systolic blood pressure (SBP) ≥180 mmHg and/or diastolic blood pressure (DBP) ≥110 mmHg despite medical therapy.
* Severe respiratory diseases (Global Initiative for Chronic Obstructive Lung Disease (GOLD) stage III-IV chronic obstructive pulmonary disease, or forced vital capacity (FVC) <50% predicted).
* Baseline bradycardia (<50) or mean arterial blood pressure less than 60mmHg.
* Emergency surgeries.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The prospective observational study will be conducted in orthopedic theatre in Cairo University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Predictive ability of the transverse diameter of the right common femoral vein (RCFV) | At end-expiration (Up to 15 minutes)
  The predictive ability of the transverse diameter of the right common femoral vein (RCFV), measured by ultrasound before spinal anesthesia, for the development of post-spinal hypotension in geriatric patients undergoing orthopedic surgery.

SECONDARY OUTCOMES:
Severity of post spinal hypotension | 24 hours postoperatively
  Severity of post spinal hypotension [defined as a decrease in the mean arterial pressure (MAP) >20% from baseline]. Severity of hypotension, classified as:
  * Mild: 20-30% decrease in MAP from baseline.
  * Moderate: 30-40% decrease in MAP from baseline.
  * Severe: >40% decrease in MAP from baseline or absolute MAP <60 mmHg.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as hypotension and/or bradycardia will be recorded.
Requirement of rescue medications | 24 hours postoperatively
  Requirement of rescue medications will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.